CLINICAL TRIAL: NCT02294838
Title: Feasibility Study of MRI Imaging on Parotid Gland Stimulation
Acronym: SPIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCCA H14-02236
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Parotid Neoplasms
MeSH Terms: conditions — Parotid Neoplasms | interventions — Magnetic Resonance Imaging; Citric Acid; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI with parotid gland stimulation (Experimental): All participants will have MRI imaging of the parotid gland with IV Gadovist pre and post parotid stimulation with lemon juice. 0.05 ml/kg of Gadovist (at 4 ml/s) and 20 ml of saline flush (also at 4 ml/s) will be administered. Approximately three minutes after scan commencement, the salivary glands will be stimulated by orally administering a small portion (≈5 ml) of Citric acid.
  Interventions: Device: MRI; Other: Citric acid; Other: Gadovist

INTERVENTIONS:
Device: MRI — Participants will undergo MR imaging of the parotid gland pre and post stimulation. Perfusion images will be acquired using a time-resolved, spoiled GE sequence with 1×1×2 mm spatial resolution, approximately one second 3D temporal resolution, and image technique/contrast parameters TR = 2.8 ms and TE = 0.9 ms.
  Other Names: Magnetic resonance imaging
Other: Citric acid — 5 mls of 2% citric Acid will be delivered to the oral cavity via a syringe and Tygon tubing at two separate time intervals in order to stimulate the parotid gland during the MRI scanning process.
Other: Gadovist — Upon commencement of the scan, 0.05 ml/kg of Gadovist (at 4 ml/s) and 20 ml of saline flush (also at 4 ml/s) will be administered.

SUMMARY:
The aim of this study is to determine the feasibility of demonstrating the following physiologically-descriptive quantities ('metrics'): the volume of plasma/volume of tissue (νp), Apparent Diffusion Coefficient (ADC), the volume of extracellular extravascular space per volume of tissue (νe), and the contrast agent transfer coefficients (Ktrans) pre and post parotid stimulation in 10 healthy volunteers. Feasibility will be defined as 80% of volunteers achieving detectable signal changes in pre/post salivary MR images.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objective:

Feasibility will be defined as 80% of volunteers achieving detectable signal changes in pre/post salivary MR images (in either the IVIM or the DCE scans).

BACKGROUND INFORMATION AND RATIONALE

It is well known that loss of salivary function in the parotid glands leads to an elevated risk of chronically dry-mouth. Xerostomia is thought to result from salivary function loss due to damage of the functional aspects of the (saliva-producing) parotid gland, but the precise nature is unknown. Recent reports have found regional dose susceptibility in rat parotid(1); delivering dose to one region of the parotid results in a different incidence of xerostomia than would that same dose to another region. Similarly, regional dose susceptibility of subjective xerostomia (i.e. patient-reported) has been noted in human parotid(2). It is presently unclear to what extent these findings relate to objective functional loss, recovery, or xerostomia in humans. With this motivation, the investigators launched a preliminary project to search for changes of parotid salivary function resulting from irradiation during treatment for head-and-neck cancers. The Investigators hypothesis was that certain regions of the parotid are more susceptible to radiation damage than others.

To test this hypothesis, data collected prospectively from one-hundred patients who underwent head-and-neck cancer treatment was analyzed for correlation between regional dose and salivary function response. Three-dimensional dose distributions were harvested from patient dose data and organ contours sub- segmented into a variety of regional "pieces". Sub-segmentation was guided by clinical recommendation. Saliva output collected by clinical staff was compared before and after treatment to provide a quantitative means of establishing salivary response. The investigators were able to demonstrate salivary function loss and recovery, but were unable to demonstrate regional susceptibility.

It was found that simple (scalar) saliva measurements and anatomical information alone do not provide enough information for the functional biology that the investigators are trying to describe. To investigate methods of obtaining functional data, the investigators have engaged with Dr Stefan Reinsberg - a researcher in the Department of Physics and Astronomy at the UBC. He develops methods for clinical and preclinical MRI for the diagnosis, planning and treatment monitoring of cancer. Techniques of particular interest to him are dynamic contrast-enhanced MRI and diffusion-weighted imaging. Through advanced statistical means he attempts to maximize the information obtained about the functional status of tissue under investigation.

As the precise site of radiation damage is thought to be the functional components (i.e., parenchyma) of the parotid, it is our belief that the use of patient-specific three dimensional anatomical and functional information is the key to understanding. Therefore, our previous data collection will be used to augment a non-invasive technique, known as Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI), which will allow us to precisely quantify regional gland function while also providing a clearer view of the glandular anatomy.

This data will be collected to optimize the technique and as preliminary (proof of concept) for an intended future protocol that will be performed on head-and-neck Intensity-Modulated Radiotherapy Treatment patients at three instances: prior to radiotherapy, and both three months and one year after conclusion of the treatment.

TRIAL DESIGN Sample size 10, proof of concept feasibility trial where preliminary data can be utilized for future study in patients undergoing active radiotherapy.

ELIGIBILITY CRITERIA There will be NO EXCEPTIONS to eligibility requirements at the time of registration. Questions about eligibility criteria should be addressed PRIOR to registration.

The eligibility criteria for this study have been carefully considered. Eligibility criteria are standards used to ensure that patients who enter this study are medically appropriate candidates for this therapy. For the safety of the participants, as well as to ensure that the results of this study can be useful for making treatment decisions regarding other patients with similar diseases, it is important that no exceptions be made to these criteria for admission to the study.

Participants must fulfill all of the following criteria to be eligible for admission to the study:

Age ≥ 18 Healthy normal volunteer

INELIGIBILITY CRITERIA

Subjects who fulfill any of the following criteria are not eligible for admission to the study:

Pregnant women Scheduled to take unusual or uncommon chemotherapy agents or medication Previous or about to undertake a course of radiotherapy Previous surgery to neck such as a lymph node dissection. Must not have, or be willing to replace, metal fillings or other foreign objects which will seriously impede image collection or analysis.

No contraindication to an MRI

PRE- MRI EVALUATION

Biochemistry Creatinine (GFR) <100 Dental assessment Check MRI check list to ensure suitability

REGISTRATION PROCEDURES

ENTRY PROCEDURES A reason for ineligibility will be recorded for all participants that are screened for the study but found to be ineligible. A record will be kept of all eligible participants that decline participation.

TRIAL PROCEDURES

MRI scans will take place at the University of British Columbia Vancouver. Tissue relaxation constant (T1) and magnetization value (M0) maps will be derived from 3 spoiled gradient echo (GE) images acquired with flip angles α = 2◦, 10◦, and 30◦, 1×1×2 mm spatial resolution, and image technique/contrast parameters TR = 2.8 ms and TE = 0.9 ms. T1 and M0 maps will be computed using image data using an L-M fitting algorithm according to the steady state signal equation.

Perfusion images will be acquired using a time-resolved, spoiled GE sequence with 1×1×2 mm spatial resolution, approximately one second 3D temporal resolution, and image technique/contrast parameters TR = 2.8 ms and TE = 0.9 ms. Upon commencement of the scan, 0.05 ml/kg of Gadovist (at 4 ml/s) and 20 ml of saline flush (also at 4 ml/s) will be administered. Approximately three minutes after scan commencement, the salivary glands will be stimulated by orally administering a small portion (≈5 ml) of lemon juice. Total perfusion scan time is expected to be 10 minutes, and the superior/inferior scan length will chosen to encompass both the parotid and submandibular glands.

Time dependent concentration maps will be derived from perfusion images and both pre-contrast T1 and M0 maps. An "extended Kety"-type model will be fit to the data with the intent of extracting the following physiologically-descriptive quantities ('metrics'): the volume of plasma/volume of tissue (νp), Apparent Diffusion Coefficient (ADC), the volume of extracellular extravascular space per volume of tissue (νe), and the contrast agent transfer coefficients (Ktrans).

Equipment 2% citric Acid will be delivered to the oral cavity via a syringe and Tygon tubing at two separate time intervals in order to stimulate the parotid gland.

EVALUATION DURING AND AFTER PROTOCOL TREATMENT

A trained medical personnel will be present during the MRI procedure to ensure patient safety is maintained through out. After the scan is completed the volunteer will not be required to attend any further follow up appointments.

ADVERSE EVENTS

Definition of a Reportable Serious Adverse Event

All serious adverse events which are unexpected and related to protocol Investigation must be reported in an expedited manner (see Section 11.2 for reporting instructions). These include events occurring during the MRI scan (until 30 days after) and at any time afterwards.

Unexpected adverse events are those which are not consistent in either nature or severity with information contained in the product monograph or package insert.

Adverse events considered related to protocol investigation are those for which a relationship to the protocol investigation cannot reasonably be ruled out.

A serious adverse event (SAE) is any adverse event that: results in death, is life-threatening,requires inpatient hospitalization or prolongation of existing hospitalization (excluding hospital admissions for study drug administration, transfusions, scheduled elective surgery and admissions for palliative or terminal care),results in persistent or significant disability or incapacity or is a congenital anomaly/birth defect Medical and scientific judgement should be exercised in deciding whether expedited reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the events listed above.

Serious Adverse Event Reporting Instructions

All reportable serious adverse events must be reported within 3 days to the Research Ethics Board.

PROTOCOL DISCONTINUATION

Criteria for Discontinuing Protocol Treatment

participants may stop protocol if: Intercurrent illness Unacceptable toxicity as defined in Section 14.4 Request by the subject

Safety Monitoring Adverse events to the contrast agent (Gadovist) will be monitored on an ongoing basis by the study team.

Any grade 5 toxicity (death) that is possibly, probably or definitely caused by the contrast agent will result in suspension of accrual and investigation by the investigator team.

Any life threatening reactions or Nephrogenic Systemic fibrosis will result in suspension of accrual and investigation by the investigator team.

Although the images will not be formally reviewed by a radiologist, it is possible that the imaging may identify unexpected abnormalities. The participants will not be issued with a diagnostic report however if an abnormality is detected, the participants and their general practitioner (with the participants permission) will be informed so that further investigations and appropriate referral can be made.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 Healthy normal volunteer

Exclusion Criteria:

Pregnant women Scheduled to take unusual or uncommon chemotherapy agents or medication Previous or about to undertake a course of radiotherapy Previous surgery to neck such as a lymph node dissection. Must not have, or be willing to replace, metal fillings or other foreign objects which will seriously impede image collection or analysis.

No contraindication to an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility study of MRI imaging on parotid gland stimulation. | time to recruit 10 healthy volunteers (approximately 4 months)
  Feasibility will be defined as 80% of volunteers achieving detectable signal changes in pre/post salivary stimulation MR images. The following physiologically-descriptive quantities ('metrics') will be measured: the volume of plasma/volume of tissue (νp), Apparent Diffusion Coefficient (ADC), the volume of extracellular extravascular space per volume of tissue (νe), and the contrast agent transfer coefficients (Ktrans) pre and post parotid stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonn Wu, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] van Luijk P, Faber H, Schippers JM, Brandenburg S, Langendijk JA, Meertens H, Coppes RP. Bath and shower effects in the rat parotid gland explain increased relative risk of parotid gland dysfunction after intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2009 Jul 15;74(4):1002-5. doi: 10.1016/j.ijrobp.2009.03.039. PMID 19545785
- [Background] Buettner F, Miah AB, Gulliford SL, Hall E, Harrington KJ, Webb S, Partridge M, Nutting CM. Novel approaches to improve the therapeutic index of head and neck radiotherapy: an analysis of data from the PARSPORT randomised phase III trial. Radiother Oncol. 2012 Apr;103(1):82-7. doi: 10.1016/j.radonc.2012.02.006. Epub 2012 Mar 21. PMID 22444242